CLINICAL TRIAL: NCT06156150
Title: The Role and Mechanism of B7-H4/ATF3 Axis From Glioma Associated Macrophages in Treatment Resistance of Cancer Vaccine
Brief Title: The Role of B7-H4 in Tumor Vaccine
Status: Recruiting | Type: Observational
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Yu Yao, MD, Professor, Huashan Hospital
Other Study IDs: KY2023-997; 8230162487 (Other Grant/Funding Number: The National Natural Science Foundation of China)
Record Dates: First submitted 2023-11-26; First posted 2023-12-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Glioma
Keywords: glioma; treatment resistance; immunotherapy; cancer vaccine; macrophage
MeSH Terms: conditions — Glioma | interventions — Cancer Vaccines

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- glioma patients receiving conventional treatment: surgery+radiotherapy+chemotherapy
- glioma patients with tumor vaccine: surgery+radiotherapy+chemotherapy+tumor vaccine
  Interventions: Biological: tumor vaccine

INTERVENTIONS:
Biological: tumor vaccine — DC vaccine produced by the Team
  Groups: glioma patients with tumor vaccine

SUMMARY:
Glioma patients have poor prognosis because of limited choices of treatment. Therapeutic cancer vaccines have been proved to improve survival in glioma, but resistance is a new challenge for vaccine treatment, and the mechanism is unclear. The applicant found in previous papers that glioma cells induced B7-H4 overexpression in macrophages, and the expression level of B7-H4 is highly correlated with vaccine resistance. Preliminary experiments indicated that B7-H4 protein in macrophages inhibited the expression of ATF3, STAT1 and CXCL9/10, which also resulted in decreased T cell infiltration in glioma model of mouse and was a negative factor of vaccine benefits. Therefore, the applicant hypothesize that B7-H4 inhibits STAT1 transcription by reducing expression of ATF3, resulting in decreased phosphorylated-STAT1 in nucleus, which inhibiting expression and secretion of chemokines 9/10. Thereby, reduced infiltration of T cells in microenvironment will be followed, which ultimately promotes resistance of vaccine treatment in glioma. The follow-up plan of this project will be conducted based on the cells, organoid platform and animal experiments to confirm the role and mechanism of macrophage-derived B7-H4 in secretion of chemokines for T cells and treatment resistance of vaccines. Moreover, the DC vaccine produced by team of the applicant will be used to assess the probability of reversing vaccine resistance when intervening B7-H4 axis. Finally, a model for evaluating clinical benefits from vaccine will be established based on data from clinical trials combining with expression of B7-H4 and clinicopathologic features. This study will provide new evidences for the treatment of cancer vaccines in gliomas.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

The patients with glioma in the Department of Neurosurgery of Huashan Hospital Affiliated to Fudan University who meet the following three conditions can be enrolled

1. They were 18-80 years old, male and female;
2. The pathological results of frozen section during operation were gliomas;
3. Tissue (6 mm * 6 mm) can be used for cell sorting on the basis of not affecting clinical routine diagnosis;
4. Sign informed consent.

Exclusion Criteria:

Patients who meet any of the following criteria will not be included in this study:

1. Participants in other clinical trials;
2. Pregnant women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing glioma surgery at Huashan Hospital
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2023-11-26 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
IHC analysis | 36 months
  Different expression level of proteins (CD3,CD8,B7-H4 et.ac) in Gliomas with different grades and molecular subgroups (100 cases) will be measured using immunohistochemical.

SECONDARY OUTCOMES:
Transcriptomics | 36 months
  The issues collected will be used for transcriptome sequencing to measure gene expression level.
Immunomics | 36 months
  The issues collected will be used for TCR/BCR sequencing to measure clonality of lymphocytes
Proteomics | 36 months
  The issues collected will be used for proteomic sequencing to measure gene expression level in protein
Radiomics | 36 months
  The features from images will be extracted using algorithm of Deep-learning or Radiomics
Genomics | 36 months
  The issues collected will be used for whole genome sequencing or whole exome sequencing to measure gene mutations.

CONTACTS AND LOCATIONS:
Locations (1):
- Di Chen, Shanghai, Shanghai Municipality, China